CLINICAL TRIAL: NCT02867137
Title: Diagnostic Potential of S100B and GFAP in Prehospital Rule-out of Intracranial Lesions in Patients Suffering Mild Traumatic Brain Injury (TBI)
Brief Title: Biomarkers in Prehospital Rule-out of Intracranial Lesions in TBI Patients
Acronym: PreTBI I
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Protokol_v2_270616_PreTBI_I
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mild TBI patients
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling from peripheral venous catheter routinely inserted in trauma patients during transportation

SUMMARY:
The PreTBI I study will investigate whether prehospital blood samples drawn already in the ambulance can rule-out intracranial lesions in patients suffering head trauma. The study aims to improve triage and treatment of patients suffering mild head trauma, who are considered low-risk patients. These patients do not always benefit from hospitalization, but are nevertheless admitted on precaution, as clinical assesment can be difficult.

Hypotheses:

1. A prehospital measurement of serum S100B ≤ 0,10 microgram/L in mild TBI patients rules out traumatic intracranial lesion with a sensitivity >97%.
2. A prehospital measurement of serum GFAP (glial acidic fibrillary protein) in mild TBI patients rules out traumatic intracranial lesion with sensitivity >97% and results in lower false positive rate than S100B.
3. Prehospital measurements of both GFAP and S100B results in lower false positive rates than in-hospital measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with Glasgow Coma Score (GCS) ≥13-15 and a loss of consciousness for less than 30 min and/or alteration of mental state (being dazed, confused or disorientated) and/or loss of memory for events immediately before and/or after the trauma. The emergency medical service staff will be guided through the inclusion and consent procedures by a simple tablet algorithm.

Exclusion Criteria:

* Patients <18 years, GCS <13, >6 hours elapsed after trauma, unknown time of trauma, multi trauma, known dementia, chronic psychosis or active central nervous system pathology.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years) suffering isolated head trauma and receiving an ambulance dispatched by the prehospital emergency medical services in the Central Denmark Region.
Sampling Method: Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of se-S100B in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.
Specificity of se-S100B in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.
Positive predictive value of se-S100B in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.
Negative predictive value of se-S100B in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.

SECONDARY OUTCOMES:
Sensitivity of se-GFAP in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.
Specificity of se-GFAP in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.
Positive predictive value of se-GFAP in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.
Negative predictive value of se-GFAP in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
  Intracranial lesion comprises abnormal CTC (Marshall Computed Tomography Classification) and/or neurosurgical observation/intervention being death <7 days secondary to head injury or the need of following procedures: craniotomy, elevation of skull fracture, intracranial pressure monitoring or intubation for head injury. Abnormal CTC findings comprise any type of intracranial haemorrhage including subdural, epidural, subarachnoid, intracerebral haemorrhage, edema, pneumocephalus, cerebral contusion or skull cap/base fractures.

OTHER OUTCOMES:
Biomarker dynamics between prehospital and in-hospital se-S100B in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
Biomarker dynamics between prehospital and in-hospital se-GFAP in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma
Biomarker dynamics between prehospital and in-hospital combination of se-S100B andse-GFAP values in relation to a binary outcome of clinical patient outcome measured by a yes/no question of "intracranial lesion" pick yes/no | in relation to event within 7 days of trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital Emergency Medical Services, Central Denmark Region, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seidenfaden SC, Kjerulff JL, Juul N, Kirkegaard H, Moller MF, Munster AB, Botker MT. Diagnostic accuracy of prehospital serum S100B and GFAP in patients with mild traumatic brain injury: a prospective observational multicenter cohort study - "the PreTBI I study". Scand J Trauma Resusc Emerg Med. 2021 Jun 2;29(1):75. doi: 10.1186/s13049-021-00891-5. PMID 34078435